CLINICAL TRIAL: NCT04249791
Title: Feasibility Assessment of Assisted Laparoscopic-robotic Hysterectomy for Uterine Transplantation in Live-donor Patient. Description of the Donor and Recipient Surgical Technique.
Brief Title: Laparoscopic-robotic Hysterectomy for Uterine Transplantation in Live-donor Patient.
Acronym: transplant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Barretos Cancer Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uterine Transplant
Record Dates: First submitted 2020-01-07; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2019-08

CONDITIONS: Uterine Anomaly
Keywords: uterine transplant; robotic surgery; donor; recipient; uterine anomaly
MeSH Terms: conditions — Uterine Anomalies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Uterus Transplantation (Experimental): Patients undergo transplantation of the uterus from live donor.
  Interventions: Procedure: Transplantation of the uterus from live donor.

INTERVENTIONS:
Procedure: Transplantation of the uterus from live donor. — Laparoscopic-robotic hysterectomy for uterine transplantation in live-donor patient.

SUMMARY:
Currently, there is no standard and indicated standard access route for uterine removal in the uterine transplant donor patient. The aim of the study is to show the feasibility of performing this procedure by replicating in our center the results found in other recent studies and to try to reduce the surgery time for both the donor and recipient patients.

DETAILED DESCRIPTION:
Few cases have been performed worldwide by laparotomic and, more recently, laparoscopic and assisted robotic access pathways. This is a clinical trial with 6 participants (3 donors and 3 recipients) to investigate the feasibility of an assisted laparoscopic-robotic surgical access route for uterine removal in the donor patient in uterine transplants. In the receiving patient, conventional surgery (midline incision) will be performed for uterine transplantation and vascular anastomoses.

ELIGIBILITY:
Inclusion Criteria:

* Desire for uterine transplantation as a donor of the uterus (with family relationship with the donor patient);
* At least one pregnancy before

Exclusion Criteria:

* comorbidities that contraindicate a surgical procedure
* Women who do not understand the study;
* Women subject to the regime that determines significant vulnerability to the participant (eg prisoners, indigenous, etc.)
* ABO blood test mismatch between donor and recipient patient.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-06-25 (Estimated); Study Completion 2021-06-25 (Estimated)

PRIMARY OUTCOMES:
transplant sucess rate | 2 years after transplantation
  Assessed by records from Barretos Cancer Hospital

SECONDARY OUTCOMES:
Live births after uterus transplantion | 2 years after transplantation
  Assessed by records from Barretos Cancer Hospital
Pregnancy rate | 2 years after transplantation
  Assessed by records from Barretos Cancer Hospital

CONTACTS AND LOCATIONS:
Overall Officials: MARCELO DE A VIEIRA, MD, Principal Investigator — Barretos Cancer Hospital
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil

REFERENCES:
- [Derived] Vieira MA, Souza C, Nobrega L, Reis R, Andrade C, Schmidt R, Carvalho L. Uterine Transplantation with Robot-assisted Uterus Retrieval from Living Donor: First Case in Brazil. J Minim Invasive Gynecol. 2021 Nov;28(11):1817. doi: 10.1016/j.jmig.2021.08.028. Epub 2021 Sep 4. PMID 34487890